CLINICAL TRIAL: NCT03148886
Title: Advanced Breast Cancer and Lifestyle Exercise Study
Acronym: ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Claude Bernard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABLE
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Breastcancer
Keywords: Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PA intervention (Experimental): The intervention consisted in a home-based adapted PA program defined at the inclusion, according to patient's capacities.
  Interventions: Other: PA intervention

INTERVENTIONS:
Other: PA intervention — The program is individualized according to age, fitness level, place of residence, access to adapted specific training group or associations, PA preferences and wishes of each participant. Patients are informed of the recommendations in terms of PA, and the target of 150min per week in order to maintain health benefits. Patients are asked to walk at least 30 minutes per day and increase their activities into daily routine. Several individual strategies are established with the patients to attain their objectives and increase their daily life PA.
  Withings® PA trackers have been used to provide an incentive effect to increase PA, to measure the number of steps per day and make people think about their PA. Patients wore a Withings Go® wristband PA tracker throughout the whole study and had in real time a feedback on their number of steps per day.
  A 7 mL blood sample is collected at baseline (D1) and at the end of the 6-month study (M6) for the biological study.

SUMMARY:
About 5% of breast cancers are metastatic at diagnosis and 20-30% of localized breast cancer become secondarily metastatic.Thanks to recent therapeutic advances, the median survival ranges between 12 months in 1970 and 18 to 24 months in 2000. However, patients suffer from many detrimental symptoms such as fatigue, pain related to treatment and metastasis. The physical, biological, psychological and clinical benefits of physical activity (PA) during treatment in patients with localized breast cancer have been widely demonstrated. Numerous studies investigated the effect of PA in non-metastatic breast cancer, but to our knowledge, only four interventional studies worldwide focused on the implementation of PA in patients with metastatic breast cancer.It seems appropriate to investigate the feasibility of PA intervention with patients with metastatic breast cancer to see if the observed effects in localized breast cancer are confirmed in metastatic breast cancer population. The ABLE study is an interventional cohort designed to assess the feasibility of a 6-month adapted physical activity intervention, performed under real life conditions in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 78 years old,
* newly diagnosed with a metastatic breast cancer (i.e. within the last 3 months)
* treated in the CLB by chemotherapy, and/or radiotherapy and/or hormonotherapy and/or targeted therapy.
* ECOG Performance status <2,
* being French-speaking
* able to complete questionnaires and follow instructions in French
* valid health insurance affiliation.
* medical certificate of no contraindications to exercise physical activity

Exclusion Criteria:

* untreated brain metastases
* uncontrolled cardiac disease,
* contraindications to PA,
* unable to be followed for medical, social, familial, geographical or psychological reasons over the study duration,
* deprivation of liberty by court or administrative decision
* pregnancy

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving the physical activity program recommendations | 6 months
  150 min per week of moderate PA assessed by the IPAQ

SECONDARY OUTCOMES:
Variation of oxidative stress | 6 months
  7mL blood sample is collected at baseline and at the end of the study
Investigate the effects of a PA intervention on fitness level | 6 months
  IPAQ in MET-min per week
Investigate the effects of a PA intervention on fitness level | 6 months
  6-min walk test in meters
Investigate the effects of a PA intervention on fitness level | 6 months
  VO2 peak in ml per kg per minute
Investigate the effects of a PA intervention on fitness level | 6 months
  strength test in kilograms
Investigate the effects of a PA intervention on quality of life | 6 months
  EORTC QLQ-C30
Investigate the effects of a PA intervention on quality of life | 6 months
  BR-23
Investigate the effects of a PA intervention on fatigue | 6 months
  PIPER scale
Investigate the effects of a PA intervention on social deprivation | 6 months
  EPICES score
Investigate the barriers and facilitators of adherence to a PA program | 6 months
  Specific questionnaire
Investigate the effects of a PA intervention on changes in anthropometrics | 6 months
  BMI in kilograms per m²
Investigate the effects of a PA intervention on changes in anthropometrics | 6 months
  waist circumference in centimeters
Investigate the effects of a PA intervention on changes in anthropometrics | 6 months
  Weight in kilograms
Investigate the effects of a PA intervention on changes in anthropometrics | 6 months
  Hip circumference in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delrieu L, Touillaud M, Perol O, Morelle M, Martin A, Friedenreich CM, Mury P, Dufresne A, Bachelot T, Heudel PE, Fervers B, Tredan O, Pialoux V. Impact of Physical Activity on Oxidative Stress Markers in Patients with Metastatic Breast Cancer. Oxid Med Cell Longev. 2021 Jul 16;2021:6694594. doi: 10.1155/2021/6694594. eCollection 2021. PMID 34326920
- [Derived] Delrieu L, Pialoux V, Perol O, Morelle M, Martin A, Friedenreich C, Febvey-Combes O, Perol D, Belladame E, Clemencon M, Roitmann E, Dufresne A, Bachelot T, Heudel PE, Touillaud M, Tredan O, Fervers B. Feasibility and Health Benefits of an Individualized Physical Activity Intervention in Women With Metastatic Breast Cancer: Intervention Study. JMIR Mhealth Uhealth. 2020 Jan 28;8(1):e12306. doi: 10.2196/12306. PMID 32012082
- [Derived] Delrieu L, Vallance JK, Morelle M, Fervers B, Pialoux V, Friedenreich C, Dufresne A, Bachelot T, Heudel PE, Tredan O, Perol O, Touillaud M. Physical activity preferences before and after participation in a 6-month physical activity intervention among women with metastatic breast cancer. Eur J Cancer Care (Engl). 2020 Jan;29(1):e13169. doi: 10.1111/ecc.13169. Epub 2019 Sep 30. PMID 31571315
- [Derived] Delrieu L, Perol O, Fervers B, Friedenreich C, Vallance J, Febvey-Combes O, Perol D, Canada B, Roitmann E, Dufresne A, Bachelot T, Heudel PE, Tredan O, Touillaud M, Pialoux V. A Personalized Physical Activity Program With Activity Trackers and a Mobile Phone App for Patients With Metastatic Breast Cancer: Protocol for a Single-Arm Feasibility Trial. JMIR Res Protoc. 2018 Aug 30;7(8):e10487. doi: 10.2196/10487. PMID 30166274